CLINICAL TRIAL: NCT06236347
Title: Scale and Evaluate Smoking Cessation and COPD Screening E-Visits to Rural Health Clinics
Brief Title: Rural COPD E-Visit Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Jennifer Dahne, Associate Professor - Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00132325; 6 U66RH31458-05-01 (Other Grant/Funding Number: Telehealth Center of Excellence)
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Smoking cessation electronic visit (e-visit) (Experimental): This group will be sent 1) an invitation to complete an electronic visit (e-visit) focused on cigarette smoking and 2) an invitation to complete a follow-up e-visit one-month after the initial e-visit.
  Interventions: Behavioral: Smoking cessation e-visit
- Treatment as usual (TAU) (Active Comparator): This group will be provided information about the state quitline and about the importance of quitting smoking and it will be recommended that they contact their PCP to schedule a medical visit to discuss quitting smoking.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Smoking cessation e-visit — Electronic visits (e-visits) for smoking cessation
  Arms: Smoking cessation electronic visit (e-visit)
Behavioral: Treatment as usual — Information about the state quitline and about the importance of quitting smoking and a recommendation to contact one's PCP to schedule a medical visit to discuss quitting smoking.
  Arms: Treatment as usual (TAU)

SUMMARY:
The purpose of this study is to evaluate an electronic visit (e-visit) for COPD screening and for quitting smoking. Participants will be randomly assigned to receive either the smoking cessation e-visit or not. The e-visit will look similar to an online questionnaire asking about smoking history, preferences for cessation medications, and chronic COPD symptoms. Participants may receive a prescription for a smoking cessation medication as an outcome of the e-visit, if randomized to the e-visit group, but there is no requirement to take any medication. This study consists of questionnaires and breath samples provided at 4 separate time points throughout the study. Participation in this study will take about 24 weeks.

DETAILED DESCRIPTION:
More than 16 million Americans have COPD and millions more suffer from COPD but have not yet been diagnosed or treated1. COPD is now concentrated within rural communities and those who reside in rural areas as compared to those who reside in large metropolitan areas have both higher COPD incidence (8% vs. 5%) and higher COPD-related death rates (55 per 100,000 vs. 32 per 100,000)2. Telehealth strategies to implement evidence-based best practice for COPD may be particularly impactful among rural communities as such treatment modalities can extend the reach of traditional COPD prevention, diagnosis, and treatment strategies.

In light of the significant public health impact of COPD, the National Heart Lung, and Blood Institute (NHLBI) issued a COPD National Action Plan in 2017. A key goal within this national action plan is to improve the diagnosis, prevention, treatment, and management of COPD by improving the quality of care delivered across the health care continuum. Because COPD is most commonly caused by cigarette smoking, investigators focus work herein on COPD early detection among cigarette smokers and on leveraging telehealth to extend the reach of evidence-based smoking cessation treatment (i.e., medications and counseling for smoking cessation) for those at risk for COPD. This work will build upon and extend our team's ongoing efforts to develop a smoking cessation electronic visit (e-visit) that can be proactively delivered to all adult MUSC patients who have been identified via the electronic health record as cigarette smokers. E-visits are embedded into the most common electronic health record (EHR) systems (e.g., Epic, Allscripts, and others) and offer a secure platform through which patients can remotely supply providers with health information. Providers in turn can deliver personalized instructions and/or treatment to the patient. Herein, investigators will leverage this proactive, scalable platform to: 1) deliver smoking cessation treatment to adults at risk for COPD and 2) improve rates of COPD early detection and accurate diagnosis. The ultimate goal of this line of work is to improve the quality of care and associated outcomes among patients at risk for COPD. investigators focus specifically on residents of rural areas given considerably higher smoking prevalence in the most rural parts of South Carolina.

ELIGIBILITY:
Inclusion criteria:

* Current cigarette smoking, defined as smoking 1+ cigarettes per day, for 20+ days out of the last 30, for the last 6+ months
* Age 40+
* Enrolled in Epic's MyChart program or willing to enroll
* Possess a valid e-mail address that is checked daily to access study assessments and MyChart messages
* Owner of an iOS or Android compatible smartphone to provide remote CO readings
* Have a valid address at which mail can be received (for mailing iCO™)
* English fluency

Exclusion criteria:

* COPD on their problem list within Epic or prior diagnosis of COPD noted elsewhere within the EHR

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Smoking Cessation | Month 1
  Self-reported smoking via Timeline Follow Back will be biochemically verified via breath CO, with abstinence defined as CO of ≤ 4 ppm. Self-report and CO data will be utilized together to determine 7-day PPA.
Smoking Cessation | Month 3
  Self-reported smoking via Timeline Follow Back will be biochemically verified via breath CO, with abstinence defined as CO of ≤ 4 ppm. Self-report and CO data will be utilized together to determine 7-day PPA.
Smoking Cessation | Month 6
  Self-reported smoking via Timeline Follow Back will be biochemically verified via breath CO, with abstinence defined as CO of ≤ 4 ppm. Self-report and CO data will be utilized together to determine 7-day PPA.
Reduction in Cigarettes Per Day | Month 1
  Reduction in cigarettes per day of 50% via self-report timeline follow back assessment.
Reduction in Cigarettes Per Day | Month 3
  Reduction in cigarettes per day of 50% via self-report timeline follow back assessment.
Reduction in Cigarettes Per Day | Month 6
  Reduction in cigarettes per day of 50% via self-report timeline follow back assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States